CLINICAL TRIAL: NCT04290312
Title: Absorption and Bioavailability of Major Monoterpenes in Mastiha Oil; a Kinetic Study in Humans.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harokopio University (Other)
Responsible Party: Principal Investigator, Andriana C Kaliora, Assistant Professor in Foods and Human Nutrition, Harokopio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MASTIHA OIL-BIO-GR
Record Dates: First submitted 2020-02-24; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Absorption
Keywords: mastiha oil, bioavailability
MeSH Terms: interventions — mastiha

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mastiha oil (Other): As a control to the experimental design, timepoint 0 was considered.
  Interventions: Other: Mastiha oil

INTERVENTIONS:
Other: Mastiha oil — After overnight fasting, the authorized study staff inserted a plastic cannula in an arm vein of the volunteers in order to minimize discomfort during consecutive blood sampling. A blood sample was collected on time point 0h and then the volunteers consumed 1mL of MO. The dose selection was based on the study of Papada et al. (2017) who administered healthy volunteers with 10g of Mastiha (containing ~10% MO). Afterwards blood samples were collected on time points 0.5h, 1h, 2h, 4h, 6h and 24h after MO intake, and were centrifuged at 3000rpm for 10 minutes at 4◦C for plasma and serum isolation. All samples were stored at -80◦C until further analysis.

SUMMARY:
Plant derived foods contain large quantities of non-nutrient phytochemicals that have been extensively studied for their beneficial health effects on the prevention of chronic diseases. Although research on their health effects is abundant, our knowledge on absorption and bioavailability is yet narrow and in some cases zero. The concept of bioavailability involves the identification of the fraction of administered compounds that can reach plasma and body tissues in an unchanged form. The bioactivity of components in foods that are part of our nutrition, either as parent foods or as food supplements, is directly related to bioavailability, the latter being a necessary step to prove efficacy.

Mastiha Oil (MO) is extracted from the resin of Pistacia Lentiscus var. Chia (of the Anacardiaceae family), a concentrated source of monoterpenes (e.g., α-pinene, β-pinene, β-myrcene) and triterpenes (e.g., mastihadienonic acid, isomastihadienonic acid), and to a lesser extent of plant sterols, simple phenols and approximately 10% MO (Assimopoulou, & Papageorgiou, 2005, Paraschos et al, 2007, Kaliora, Mylona, Chiou, Petsios, & Andrikopoulos, 2004). MO is a 100% natural product used as a food additive and flavoring and it is manufactured according to the legal standards that make it suitable for human consumption. Its nutritional analysis is presented in Supplementary Table 1. A total of 90 components have been detected in MO (50% monoterpene hydrocarbons, 20% oxygenated monoterpenes, 25% sesquiterpenes). Monoterpenes seem to exhibit beneficial health effects contributing to mechanisms of inflammation and oxidative stress (Subramaniyan, 2017; Madhuri, & Naik, 2017).

Research upon the bioavailability of monoterpenes in humans is limited. Herein, we aimed at investigating the bioavailability of the main monoterpenes of MO in humans for the first time. To this end, a novel GC-MS-MS method was employed, since the tandem MS technique can help overcome matrix difficulties. Additionally, based on the existing data regarding the antioxidant activity of monoterpenes, the effect on human antioxidant capacity was evaluated applying the serum oxidisabilty assay.

.

DETAILED DESCRIPTION:
After enrolment, the volunteers will undergo a medical and dietary assessment and their health status will be evaluated through a complete blood count. On the day of the experiment and after overnight fasting, the volunteers will consume g of mastiha oil (1ml) and blood samples will be obtained on timepoints 0.5h, 1h, 2h, 4h, 6h and 24h after intake. Until timepoint 6h, they will be allowed to consume only water. After collection, the monoterpenes will be identified in plasma samples applying a GC-MS-MS technique. Additionally, oxidative stress will be evaluated through the CuSO4 technique in serum samples.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-40 years old
* BMI: 18.5-24.9 kg/m2

Exclusion Criteria:

* Obesity
* Alcohol or drug abuse
* Medication, vitamin or inorganic supplements
* Vegan or macrobiotic diet before and during the study
* Gastrointestinal diseases, such as atrophic gastritis, Inflammatory Bowel Disease, peptic ulcer or gastrointestinal cancer

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of monoterpenes | 24 hours
  The monoterpenes will be identified and quantified in plasma samples applying GC-MS-MS. Data will be presented through study completion in plasma concentration (μg/L).

CONTACTS AND LOCATIONS:
Overall Officials: Andriana Kaliora, Ass. Professor, Principal Investigator — Harokopio University
Locations (1):
- Harokopio University, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papada E, Gioxari A, Brieudes V, Amerikanou C, Halabalaki M, Skaltsounis AL, Smyrnioudis I, Kaliora AC. Bioavailability of Terpenes and Postprandial Effect on Human Antioxidant Potential. An Open-Label Study in Healthy Subjects. Mol Nutr Food Res. 2018 Feb;62(3). doi: 10.1002/mnfr.201700751. Epub 2017 Dec 29. PMID 29171157
- [Background] Abidi A, Aissani N, Sebai H, Serairi R, Kourda N, Ben Khamsa S. Protective Effect of Pistacia lentiscus Oil Against Bleomycin-Induced Lung Fibrosis and Oxidative Stress in Rat. Nutr Cancer. 2017 Apr;69(3):490-497. doi: 10.1080/01635581.2017.1283423. Epub 2017 Feb 17. PMID 28287322
- [Background] J C Furtado NA, Pirson L, Edelberg H, M Miranda L, Loira-Pastoriza C, Preat V, Larondelle Y, Andre CM. Pentacyclic Triterpene Bioavailability: An Overview of In Vitro and In Vivo Studies. Molecules. 2017 Mar 4;22(3):400. doi: 10.3390/molecules22030400. PMID 28273859
- [Background] Garcia-Villalba R, Larrosa M, Possemiers S, Tomas-Barberan FA, Espin JC. Bioavailability of phenolics from an oleuropein-rich olive (Olea europaea) leaf extract and its acute effect on plasma antioxidant status: comparison between pre- and postmenopausal women. Eur J Nutr. 2014 Jun;53(4):1015-27. doi: 10.1007/s00394-013-0604-9. Epub 2013 Oct 26. PMID 24158653
- [Background] Kanellos PT, Kaliora AC, Gioxari A, Christopoulou GO, Kalogeropoulos N, Karathanos VT. Absorption and bioavailability of antioxidant phytochemicals and increase of serum oxidation resistance in healthy subjects following supplementation with raisins. Plant Foods Hum Nutr. 2013 Dec;68(4):411-5. doi: 10.1007/s11130-013-0389-2. PMID 24114059
- [Background] Subramaniyan SD, Natarajan AK. Citral, A Monoterpene Protect Against High Glucose Induced Oxidative Injury in HepG2 Cell In Vitro-An Experimental Study. J Clin Diagn Res. 2017 Aug;11(8):BC10-BC15. doi: 10.7860/JCDR/2017/28470.10377. Epub 2017 Aug 1. PMID 28969111
- [Background] Saidi SA, Ncir M, Chaaben R, Jamoussi K, van Pelt J, Elfeki A. Liver injury following small intestinal ischemia reperfusion in rats is attenuated by Pistacia lentiscus oil: antioxidant and anti-inflammatory effects. Arch Physiol Biochem. 2017 Oct;123(4):199-205. doi: 10.1080/13813455.2017.1302961. Epub 2017 Mar 24. PMID 28338348
- [Derived] Papada E, Gioxari A, Amerikanou C, Galanis N, Kaliora AC. An Absorption and Plasma Kinetics Study of Monoterpenes Present in Mastiha Oil in Humans. Foods. 2020 Jul 30;9(8):1019. doi: 10.3390/foods9081019. PMID 32751415